CLINICAL TRIAL: NCT03755791
Title: A Randomized, Controlled Phase 3 Study of Cabozantinib (XL184) in Combination With Atezolizumab Versus Sorafenib in Subjects With Advanced Hepatocellular Carcinoma Who Have Not Received Previous Systemic Anticancer Therapy
Brief Title: Study of Cabozantinib in Combination With Atezolizumab Versus Sorafenib in Participants With Advanced Hepatocellular Carcinoma (HCC) Who Have Not Received Previous Systemic Anticancer Therapy
Acronym: COSMIC-312
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XL184-312; 2024-516479-34-00 (EU CTIS Number)
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Results first posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: liver; cancer; hepatocellular; carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasms; Carcinoma | interventions — cabozantinib; Sorafenib; atezolizumab

STUDY DESIGN:
Intervention Model Description: At least 740 eligible participants with advanced HCC will be randomized in a 2:1:1 ratio. Experimental arm (at least 370 participants) will receive cabozantinib plus atezolizumab. Control arm (at least 185 participants) will receive sorafenib. Single-agent cabozantinib arm (at least185 participants) will receive single-agent cabozantinib
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Experimental arm (Experimental): Participants with advanced HCC will receive cabozantinib 40 milligrams (mg) oral, once daily (qd) + atezolizumab 1200 mg infusion, once every 3 weeks (q3w)
  Interventions: Drug: Cabozantinib; Drug: Atezolizumab
- Control arm (Active Comparator): Participants with advanced HCC will receive sorafenib 400 mg twice a day (bid)
  Interventions: Drug: Sorafenib
- Single-Agent Cabozantinib arm (Other): Participants with advanced HCC will receive cabozantinib 60 mg qd
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — Supplied as 20-mg tablets; administered orally daily at 40 mg
  Other Names: XL184; Cabometyx®
  Arms: Experimental arm
Drug: Cabozantinib — Supplied as 60-mg tablets; administered orally once daily at 60 mg
  Other Names: XL184; Cabometyx®
  Arms: Single-Agent Cabozantinib arm
Drug: Sorafenib — Supplied as 200-mg tablets; administered orally twice daily at 400 mg
  Other Names: Nexavar®
  Arms: Control arm
Drug: Atezolizumab — Supplied as 1200 mg/20 mL (60 mg/mL) in sing-dose vials; administered as an intravenous (IV) infusion q3w
  Other Names: Tecentriq®
  Arms: Experimental arm

SUMMARY:
This Phase 3 study evaluates the safety and efficacy of cabozantinib in combination with atezolizumab versus the standard of care sorafenib in adults with advanced hepatocellular carcinoma (HCC) who have not received previous systemic anticancer therapy. A single-agent cabozantinib arm will be enrolled in which participants receive single agent cabozantinib in order to determine its contribution to the overall safety and efficacy of the combination with atezolizumab.

DETAILED DESCRIPTION:
This is a multicenter, randomized, open-label, controlled Phase 3 trial of cabozantinib in combination with atezolizumab versus sorafenib in adults with advanced HCC who have not received previous systemic anticancer therapy in the advanced HCC setting. The primary objective of this study is to evaluate the effect of cabozantinib in combination with atezolizumab on the duration of progression-free survival (PFS) and duration of overall survival (OS) versus sorafenib. The secondary objective is to evaluate the activity of single-agent cabozantinib compared with sorafenib in this patient population.

ELIGIBILITY:
Key Inclusion Criteria:

* Histological or cytological diagnosis of HCC or clinical diagnosis of HCC in cirrhotic patients by Computed Tomography (CT) or Computed Tomography (MRI) per the American Association for the Study of Liver Diseases (AASLD) 2018 or European Association for the Study of the Liver (EASL) 2018 guidelines.
* The participant has disease that is not amenable to a curative treatment approach (eg, transplant, surgery, ablation therapy) or locoregional therapy (eg, TACE).
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as determined by the Investigator.
* Barcelona Clinic Liver Cancer (BCLC) stage Category B or C.
* Child-Pugh Score of A.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Key Exclusion Criteria:

* Known fibrolamellar carcinoma, sarcomatoid HCC or mixed hepatocellular cholangiocarcinoma.
* Prior systemic anticancer therapy for advanced HCC including but not limited to chemotherapy, small molecule kinase inhibitors, and immune checkpoint inhibitors (ICIs). Participants who have received local intratumoral or arterial chemotherapy are eligible; local anticancer therapy within ≥ 28 days before randomization
* Radiation therapy for bone metastasis within 2 weeks, any other radiation therapy within 8 weeks prior to randomization.
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 8 weeks prior to randomization.
* Concomitant anticoagulation with oral anticoagulants

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 837 (Actual)
Dates: Start 2018-06-10 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2026-07-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Exelixis
Locations (245):
- United States (33):
  - Exelixis Clinical Site #208, Phoenix, Arizona
  - Exelixis Clinical Site #159, Tucson, Arizona
  - Exelixis Clinical Site #44, La Jolla, California
  - Exelixis Clinical Site #112, Los Angeles, California
  - Exelixis Clinical Site #200, Orange, California
  - Exelixis Clinical Site #2, Rialto, California
  - Exelixis Clinical Site #207, San Diego, California
  - Exelixis Clinical Site #109, San Francisco, California
  - Exelixis Clinical Site #54, San Francisco, California
  - Exelixis Clinical Site #58, Washington D.C., District of Columbia
  - Exelixis Clinical Site #191, Miami, Florida
  - Exelixis Clinical Site #4, Atlanta, Georgia
  - Exelixis Clinical Site #195, Chicago, Illinois
  - Exelixis Clinical Site #120, Chicago, Illinois
  - Exelixis Clinical Site #6, Baltimore, Maryland
  - Exelixis Clinical Site #7, Burlington, Massachusetts
  - Exelixis Clinical Site #11, Kansas City, Missouri
  - Exelixis Clinical Site #5, Kansas City, Missouri
  - Exelixis Clinical Site #8, St Louis, Missouri
  - Exelixis Clinical Site #1, Las Vegas, Nevada
  - Exelixis Clinical Site #14, New Brunswick, New Jersey
  - Exelixis Clinical Site #76, Albuquerque, New Mexico
  - Exelixis Clinical Site #12, Chapel Hill, North Carolina
  - Exelixis Clinical Site #39, Toledo, Ohio
  - Exelixis Clinical Site #176, Portland, Oregon
  - Exelixis Clinical Site #88, Philadelphia, Pennsylvania
  - Exelixis Clinical Site #144, Charleston, South Carolina
  - Exelixis Clinical Site #199, Dallas, Texas
  - Exelixis Clinical Site #154, Houston, Texas
  - Exelixis Clinical Site #19, Temple, Texas
  - Exelixis Clinical Site #13, Seattle, Washington
  - Exelixis Clinical Site #46, Seattle, Washington
  - Exelixis Clinical Site #3, Spokane, Washington
- Argentina (6):
  - Exelixis Clinical Site #217, City of Buenos Aires, Buenos Aires
  - Exelixis Clinical Site #213, City of Buenos Aires, Buenos Aires
  - Exelixis Clinical Site #216, City of Buenos Aires, Buenos Aires
  - Exelixis Clinical Site #219, Pilar, Buenos Aires
  - Exelixis Clinical Site #220, Rosario, Santa Fe Province
  - Exelixis Clinical Site #201, Rosario, Santa Fe Province
- Australia (11):
  - Exelixis Clinical Site #78, Camperdown, New South Wales
  - Exelixis Clinical Site #165, Darlinghurst, New South Wales
  - Exelixis Clinical Site #171, Kingswood, New South Wales
  - Exelixis Clinical Site #126, Kogarah, New South Wales
  - Exelixis Clinical Site #155, Westmead, New South Wales
  - Exelixis Clinical Site #142, Greenslopes, Queensland
  - Exelixis Clinical Site #17, Kurralta Park, South Australia
  - Exelixis Clinical Site #107, Box Hill, Victoria
  - Exelixis Clinical Site #166, Heidelberg, Victoria
  - Exelixis Clinical Site #72, Parkville, Victoria
  - Exelixis Clinical Site #190, Nedlands, Western Australia
- Austria (5):
  - Exelixis Clinical Site #150, Klagenfurt, Carinthia
  - Exelixis Clinical Site #137, Sankt Pölten, Lower Austria
  - Exelixis Clinical Site #198, Graz, Styria
  - Exelixis Clinical Site #64, Linz, Upper Austria
  - Exelixis Clinical Site #174, Vienna
- Belgium (7):
  - Exelixis Clinical Site #50, Brussels, California
  - Exelixis Clinical Site #65, Brussels
  - Exelixis Clinical Site #169, Edegem
  - Exelixis Clinical Site #148, Ghent
  - Exelixis Clinical Site #57, Haine-Saint-Paul
  - Exelixis Clinical Site #188, Leuven
  - Exelixis Clinical Site #102, Liège
- Brazil (12):
  - Exelixis Clinical Site #184, Salvador, Estado de Bahia
  - Exelixis Clinical Site #89, Belo Horizonte, Minas Gerais
  - Exelixis Clinical Site #98, Belo Horizonte, Minas Gerais
  - Exelixis Clinical Site #113, Curitiba, Paraná
  - Exelixis Clinical Site #203, Porto Alegre, Rio Grande do Sul
  - Exelixis Clinical Site #175, Barretos, São Paulo
  - Exelixis Clinical Site #121, Jaú, São Paulo
  - Exelixis Clinical Site #186, São Paulo, São Paulo
  - Exelixis Clinical Site #156, São Paulo, São Paulo
  - Exelixis Clinical Site #187, São Paulo, São Paulo
  - Exelixis Clinical Site #181, São Paulo, São Paulo
  - Exelixis Clinical Site #91, São Paulo
- Canada (7):
  - Exelixis Clinical Site #71, Calgary, Alberta
  - Exelixis Clinical Site #205, Edmonton, Alberta
  - Exelixis Clinical Site #34, Winnipeg, Manitoba
  - Exelixis Clinical Site #222, Halifax, Nova Scotia
  - Exelixis Clinical Site #194, Hamilton, Ontario
  - Exelixis Clinical Site #212, Ottawa, Ontario
  - Exelixis Clinical Site #85, Montreal, Quebec
- China (24):
  - Exelixis Clinical Site #233, Hefei, Anhui
  - Exelixis Clinical Site #228, Fuzhou, Fujian
  - Exelixis Clinical Site #225, Xiamen, Fujian
  - Exelixis Clinical Site #242, Guangzhou, Guangdong
  - Exelixis Clinical Site #227, Harbin, Heilongjiang
  - Exelixis Clinical Site #230, Zhengzhou, Henan
  - Exelixis Clinical Site #231, Changsha, Hunan
  - Exelixis Clinical Site #224, Changsha, Hunan
  - Exelixis Site #241, Changsha, Hunan
  - Exelixis Clinical Site #185, Nanjing, Jiangsu
  - Exelixis Clinical Site #221, Nanchang, Jiangxi
  - Exelixis Clinical Site #238, Nanchang, Jiangxi
  - Exelixis Clinical Site #234, Jiangyin, Jiansu
  - Exelixis Clinical Site #246, Changchun, Jilin
  - Exelixis Clinical Site #229, Changchun, Jilin
  - Exelixis Clinical Site #236, Shenyang, Liaoning
  - Exelixis Clinical Site #226, Linyi, Shandong
  - Exelixis Clinical Site #235, Chengdu, Sichuan
  - Exelixis Clinical Site #218, Hangzhou, Zhejiang
  - Exelixis Clinical Site #223, Hangzhou, Zhejiang
  - Exelixis Site #239, Beijing
  - Exelixis Clinical Site #237, Beijing
  - Exelixis Site #240, Shanghai
  - Exelixis Clinical Site #232, Shanghai
- Exelixis Clinical Site #130, Montería, Departamento de Córdoba, Colombia
- Czechia (4):
  - Exelixis Clinical Site #18, Hradec Králové
  - Exelixis Clinical Site #37, Olomouc
  - Exelixis Clinical Site #10, Prague
  - Exelixis Clinical Site #38, Prague
- France (14):
  - Exelixis Clinical Site #43, Amiens
  - Exelixis Clinical Site #27, Besançon
  - Exelixis Clinical Site #56, Bondy
  - Exelixis Clinical Site #29, Caen
  - Exelixis Clinical Site #48, Clichy
  - Exelixis Clinical Site #23, Grenoble
  - Exelixis Clinical Site #55, Lille
  - Exelixis Clinical Site #16, Lyon
  - Exelixis Clinical Site #31, Montbéliard
  - Exelixis Clinical Site #49, Montpellier
  - Exelixis Clinical Site #47, Nantes
  - Exelixis Clinical Site #51, Nice
  - Exelixis Clinical Site #20, Pessac
  - Exelixis Clinical Site #32, Vandœuvre-lès-Nancy
- Georgia (5):
  - Exelixis Clinical Site #69, Batumi
  - Exelixis Clinical Site #66, Tbilisi
  - Exelixis Clinical Site #68, Tbilisi
  - Exelixis Clinical Site #67, Tbilisi
  - Exelixis Clinical Site #70, Tbilisi
- Germany (4):
  - Exelixis Clinical Site #244, Frankfurt am Main, Hesse
  - Exelixis Clinical Site #210, Kassel, Hesse
  - Exelixis Clinical Site #214, Berlin
  - Exelixis Clinical Site #215, Hamburg
- Hong Kong (3):
  - Exelixis Clinical Site #146, Hong Kong
  - Exelixis Clinical Site #42, Hong Kong
  - Exelixis Clinical Site #9, Hong Kong
- Hungary (3):
  - Exelixis Clinical Site #140, Budapest
  - Exelixis Clinical Site #25, Debrecen
  - Exelixis Clinical Site #26, Szeged
- Exelixis Clinical Site #170, Dublin, Ireland
- Israel (4):
  - Exelixis Clinical Site #30, Jerusalem
  - Exelixis Clinical Site #33, Petah Tikva
  - Exelixis Clinical Site #40, Ramat Gan
  - Exelixis Clinical Site #35, Rehovot
- Italy (11):
  - Exelixis Clinical Site #163, Tricase, Lecce
  - Exelixis Clinical Site #53, Rozzano, Milano
  - Exelixis Clinical Site #158, Bologna
  - Exelixis Clinical Site #152, Brescia
  - Exelixis Clinical Site #147, Milan
  - Exelixis Clinical Site #149, Napoli
  - Exelixis Clinical Site #131, Novara
  - Exelixis Clinical Site #167, Roma
  - Exelixis Clinical Site #177, Torino
  - Exelixis Clinical Site #182, Torino
  - Exelixis Clinical Site #243, Udine
- Mexico (7):
  - Exelixis Clinical Site #141, Tuxtla Gutiérrez, Chiapas
  - Exelixis Clinical Site #135, León, Guanajuato
  - Exelixis Clinical Site #132, Monterrey, Nuevo León
  - Exelixis Clinical Site #133, Mexico City
  - Exelixis Clinical Site #160, Mexico City
  - Exelixis Clinical Site #134, San Luis Potosí City
  - Exelixis Clinical Site #153, Veracruz
- Netherlands (4):
  - Exelixis Clinical Site #92, Maastricht, Limburg
  - Exelixis Clinical Site #52, Amsterdam, North Holland
  - Exelixis Clinical Site #84, Rotterdam, South Holland
  - Exelixis Clinical Site #36, Utrecht
- New Zealand (2):
  - Exelixis Clinical Site #60, Grafton, Auckland
  - Exelixis Clinical Site #62, Newton, Wellington Region
- Philippines (3):
  - Exelixis Clinical Site #118, Cebu City
  - Exelixis Clinical Site #117, Pasig
  - Exelixis Clinical Site #136, Quezon City
- Poland (3):
  - Exelixis Clinical Site #41, Warsaw, Masovian Voivodeship
  - Exelixis Clinical Site #24, Gdansk, Pomeranian Voivodeship
  - Exelixis Clinical Site #15, Mysłowice, Silesian Voivodeship
- Romania (5):
  - Exelixis Clinical Site #204, Cluj-Napoca, Cluj
  - Exelixis Clinical Site #211, Cluj-Napoca, Cluj
  - Exelixis Clinical Site #202, Cluj-Napoca, Cluj
  - Exelixis Clinical Site #206, Bucharest
  - Exelixis Clinical Site #209, Iași
- Russia (9):
  - Exelixis Clinical Site #74, Kislino, Kursk Oblast
  - Exelixis Clinical Site #81, Kaluga
  - Exelixis Clinical Site #95, Krasnodar
  - Exelixis Clinical Site #108, Moscow
  - Exelixis Clinical Site #101, Murmansk
  - Exelixis Clinical Site #80, Nizhny Novgorod
  - Exelixis Clinical Site #111, Saint Petersburg
  - Exelixis Clinical Site #90, Saint Petersburg
  - Exelixis Clinical Site #73, Sochi
- Singapore (3):
  - Exelixis Clinical Site #106, Singapore
  - Exelixis Clinical Site #97, Singapore
  - Exelixis Clinical Site #116, Singapore
- South Korea (11):
  - Exelixis Clinical Site #157, Goyang-si, Gyeonggi-do
  - Exelixis Clinical Site #127, Suwon, Gyeonggi-do
  - Exelixis Clinical Site #77, Busan
  - Exelixis Clinical Site #86, Busan
  - Exelixis Clinical Site #114, Busan
  - Exelixis Clinical Site #75, Incheon
  - Exelixis Clinical Site #104, Seoul
  - Exelixis Clinical Site #105, Seoul
  - Exelixis Clinical Site #99, Seoul
  - Exelixis Clinical Site #79, Seoul
  - Exelixis Clinical Site #93, Seoul
- Spain (9):
  - Exelixis Clinical Site #28, Santander, Cantabria
  - Exelixis Clinical Site #21, Majadahonda, Madrid
  - Exelixis Clinical Site #22, Majadahonda, Madrid
  - Exelixis Clinical Site #59, Pamplona, Navarre
  - Exelixis Clinical Site #103, Barcelona
  - Exelixis Clinical Site #164, Madrid
  - Exelixis Clinical Site #63, Madrid
  - Exelixis Clinical Site #168, Valencia
  - Exelixis Clinical Site #45, Zaragoza
- Switzerland (4):
  - Exelixis Clinical Site #115, Basel
  - Exelixis Clinical Site #172, Bern
  - Exelixis Clinical Site #110, Sankt Gallen
  - Exelixis Clinical Site #61, Zurich
- Taiwan (9):
  - Exelixis Clinical Site #119, Changhua
  - Exelixis Clinical Site #162, Kaohsiung City
  - Exelixis Clinical Site #161, Taichung
  - Exelixis Clinical Site #197, Tainan
  - Exelixis Clinical Site #145, Tainan
  - Exelixis Clinical Site #82, Taipei
  - Exelixis Clinical Site #128, Taipei
  - Exelixisi Clinical Site #100, Taipei
  - Exelixis Clinical Site #94, Taoyuan District
- Thailand (4):
  - Exelixis Clinical Site #96, Pathum Wan, Bangkok
  - Exelixis Clinical Site #139, Hat Yai, Changwat Songkhla
  - Exelixis Clinical Site #143, Chiang Mai
  - Exelixis Clinical Site #183, Khon Kaen
- Turkey (Türkiye) (6):
  - Exelixis Clinical Site #189, Istanbul, Instanbul
  - Exelixis Clinical Site #193, Ankara
  - Exelixis Clinical Site #178, Ankara
  - Exelixis Clinical Site #173, Edirne
  - Exelixis Clinical Site #179, Istanbul
  - Exelixis Clinical Site #180, Malatya
- Ukraine (5):
  - Exelixis Clinical Site #125, Chernivtsi
  - Exelixis Clinical Site #122, Dnipro
  - Exelixis Clinical Site #123, Kharkiv
  - Exelixis Clinical Site #124, Odesa
  - Exelixis Clinical Site #138, Uzhhorod
- United Kingdom (6):
  - Exelixis Clinical Site #83, Bristol, England
  - Exelixis Clinical Site #87, Cambridge, England
  - Exelixis Clinical Site #151, London, England
  - Exelixis Clinical Site #129, London, England
  - Exelixis Clinical Site #192, Manchester, England
  - Exelixis Clinical Site #196, Belfast, Northern Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yau T, Kaseb A, Cheng AL, Qin S, Zhu AX, Chan SL, Melkadze T, Sukeepaisarnjaroen W, Breder V, Verset G, Gane E, Borbath I, Rangel JDG, Ryoo BY, Makharadze T, Merle P, Benzaghou F, Milwee S, Wang Z, Curran D, Kelley RK, Rimassa L. Cabozantinib plus atezolizumab versus sorafenib for advanced hepatocellular carcinoma (COSMIC-312): final results of a randomised phase 3 study. Lancet Gastroenterol Hepatol. 2024 Apr;9(4):310-322. doi: 10.1016/S2468-1253(23)00454-5. Epub 2024 Feb 13. PMID 38364832
- [Derived] Kelley RK, Rimassa L, Cheng AL, Kaseb A, Qin S, Zhu AX, Chan SL, Melkadze T, Sukeepaisarnjaroen W, Breder V, Verset G, Gane E, Borbath I, Rangel JDG, Ryoo BY, Makharadze T, Merle P, Benzaghou F, Banerjee K, Hazra S, Fawcett J, Yau T. Cabozantinib plus atezolizumab versus sorafenib for advanced hepatocellular carcinoma (COSMIC-312): a multicentre, open-label, randomised, phase 3 trial. Lancet Oncol. 2022 Aug;23(8):995-1008. doi: 10.1016/S1470-2045(22)00326-6. Epub 2022 Jul 4. PMID 35798016
- [Derived] Kelley RK, W Oliver J, Hazra S, Benzaghou F, Yau T, Cheng AL, Rimassa L. Cabozantinib in combination with atezolizumab versus sorafenib in treatment-naive advanced hepatocellular carcinoma: COSMIC-312 Phase III study design. Future Oncol. 2020 Jul;16(21):1525-1536. doi: 10.2217/fon-2020-0283. Epub 2020 Jun 3. PMID 32491932

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Arm: Cabozantinib + Atezolizumab: Participants received 40 milligrams (mg) cabozantinib oral tablets once daily + 1200 mg intravenous (IV) infusion of atezolizumab once every 3 weeks for up to 38 months.
- Single-Agent Cabozantinib: Participants received 60 mg cabozantinib oral tablets once daily for up to 38 months.
- Control Arm: Sorafenib: Participants received 400 mg sorafenib oral tablets twice daily (BID) for up to 38 months.
Period: Overall Study
Arm/Group | Experimental Arm: Cabozantinib + Atezolizumab | Single-Agent Cabozantinib | Control Arm: Sorafenib
Started | 432 | 188 | 217
Received At Least 1 Dose of Study Drug | 429 | 188 | 207
Completed | 0 | 0 | 0
Not Completed | 432 | 188 | 217
Not completed — Did not receive any study treatment | 3 | 0 | 10
Not completed — Radiographic progression | 204 | 92 | 115
Not completed — Adverse Event | 140 | 60 | 51
Not completed — Lack of Efficacy | 12 | 6 | 6
Not completed — Withdrawal by Subject | 26 | 23 | 24
Not completed — Sponsor decision, | 41 | 5 | 7
Not completed — Lost to Follow-up | 1 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 2
Not completed — Other than specified | 5 | 2 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population consisted of all participants who were randomized to any of the three study treatment arms, regardless of whether they received any study treatment.
Groups:
- Experimental Arm: Cabozantinib + Atezolizumab: Participants received 40 mg cabozantinib oral tablets once daily + 1200 mg IV infusion of atezolizumab once every 3 weeks for up to 38 months.
- Control Arm: Sorafenib: Participants received 400 mg sorafenib oral tablets twice daily for up to 38 months.
- Total: Total of all reporting groups
Arm/Group | Experimental Arm: Cabozantinib + Atezolizumab | Single-Agent Cabozantinib | Control Arm: Sorafenib | Total
Number analyzed (Participants) | 432 | 188 | 217 | 837
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 234 | 97 | 112 | 443
  >=65 years | 198 | 91 | 105 | 394
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 30 | 31 | 133
  Male | 360 | 158 | 186 | 704
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 42 | 21 | 15 | 78
  Not Hispanic or Latino | 352 | 158 | 183 | 693
  Not Reported | 38 | 9 | 19 | 66
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 127 | 64 | 72 | 263
  Black/African American | 8 | 5 | 1 | 14
  White | 217 | 95 | 111 | 423
  Other than specified | 80 | 24 | 33 | 137

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) for the Experimental Arm Versus the Control Arm in the PFS Intent to Treat (PITT) Population
Description: PFS was defined as the time from randomization to the earlier of either the date of radiographic progression defined as a 20% increase in the sum of the longest diameters of target lesions, or the unequivocal appearance of new lesions, or progression of non-target disease per Blinded Independent Radiology Committee (BIRC) or the date of death due to any cause per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Time Frame: From the date of first participant randomization up to 28 months
Population: PITT population included the first 372 participants randomized to the experimental (cabozantinib + atezolizumab) arm and control (sorafenib) arm.
Measure: Median (99% Confidence Interval); unit: months
Arm/Group | Experimental Arm: Cabozantinib + Atezolizumab | Control Arm: Sorafenib
Number analyzed (Participants) | 250 | 122
months | 6.80 [5.55 to 8.34] | 4.21 [2.79 to 7.03]
Statistical Analysis 1: Comparison: Experimental Arm: Cabozantinib + Atezolizumab vs Control Arm: Sorafenib; Test type: Other; p = 0.0012, Log Rank; Hazard Ratio (HR) = 0.63, 99% CI 2-sided [0.44 to 0.91]

2. Primary Outcome: Overall Survival (OS) for the Experimental Arm Versus the Control Arm in the ITT Population
Description: OS was defined as the time from randomization to death due to any cause.
Time Frame: From the date of first participant randomization up to 36 months
Population: ITT population included all participants randomized to the experimental (cabozantinib + atezolizumab) arm and control (sorafenib) arm.
Measure: Mean (96% Confidence Interval); unit: months
Arm/Group | Experimental Arm: Cabozantinib + Atezolizumab | Control Arm: Sorafenib
Number analyzed (Participants) | 432 | 217
months | 16.46 [14.46 to 18.56] | 15.51 [12.19 to 19.98]
Statistical Analysis 1: Comparison: Experimental Arm: Cabozantinib + Atezolizumab vs Control Arm: Sorafenib; Test type: Other; p = 0.9056, Log Rank; Hazard Ratio (HR) = 0.99, 96% CI 2-sided [0.78 to 1.24]

3. Secondary Outcome: PFS for the Single-Agent Cabozantinib Arm Versus the Control Arm in the ITT Population
Description: PFS was defined as the time from randomization to the earlier of either the date of radiographic progression per BIRC or the date of death due to any cause per RECIST version 1.1.
Time Frame: From the date of first participant randomization up to 28 months
Population: ITT population included all participants randomized to the single agent cabozantinib arm and control (sorafenib) arm.
Measure: Median (99% Confidence Interval); unit: months
Arm/Group | Single-Agent Cabozantinib | Control Arm: Sorafenib
Number analyzed (Participants) | 188 | 217
months | 5.82 [5.42 to 8.18] | 4.27 [2.86 to 6.11]

ADVERSE EVENTS:
Time Frame: Up to 39 months
Description: Safety population included all randomized participants who received at least one dose of study drug.
  The participants that did not receive any medication in the Cabozantinib + Atezolizumab and the Sorafenib were not included in the safety population.
Arm/Group | Experimental Arm: Cabozantinib + Atezolizumab | Single-Agent Cabozantinib | Control Arm: Sorafenib
All-Cause Mortality (participants affected / at risk) | 307/429 | 135/188 | 141/207
Serious Adverse Events (participants affected / at risk) | 226/429 | 88/188 | 85/207
Other Adverse Events (participants affected / at risk) | 414/429 | 182/188 | 202/207
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Experimental Arm: Cabozantinib + Atezolizumab (N=429) | Single-Agent Cabozantinib (N=188) | Control Arm: Sorafenib (N=207)
Anaemia (Blood and lymphatic system disorders) | 6 | 1 | 4
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 3 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 0 | 1
Thyroiditis (Endocrine disorders) | 2 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 8 | 4 | 4
Abdominal pain upper (Gastrointestinal disorders) | 4 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 15 | 3 | 3
Colitis (Gastrointestinal disorders) | 4 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 9 | 4 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0
Enterovesical fistula (Gastrointestinal disorders) | 0 | 0 | 1
Gastric perforation (Gastrointestinal disorders) | 0 | 1 | 0
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 3 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 1
Haemoperitoneum (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 4 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 1
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 4 | 2 | 2
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 2 | 0
Varices oesophageal (Gastrointestinal disorders) | 4 | 1 | 2
Visceral venous thrombosis (Gastrointestinal disorders) | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 5 | 3 | 1
Abscess sterile (General disorders) | 0 | 1 | 0
Asthenia (General disorders) | 7 | 2 | 2
Chest pain (General disorders) | 3 | 0 | 0
Death (General disorders) | 4 | 0 | 1
Fatigue (General disorders) | 2 | 2 | 1
General physical health deterioration (General disorders) | 5 | 1 | 2
Generalised oedema (General disorders) | 0 | 1 | 0
Inflammation (General disorders) | 1 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 2 | 0 | 1
Mucosal inflammation (General disorders) | 1 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 4 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 11 | 1 | 1
Sudden death (General disorders) | 1 | 0 | 1
Acute hepatic failure (Hepatobiliary disorders) | 0 | 2 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 2 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 1 | 1 | 0
Biloma (Hepatobiliary disorders) | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Chronic hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0
Gallbladder obstruction (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 2 | 2 | 0
Hepatic failure (Hepatobiliary disorders) | 8 | 4 | 2
Hepatitis (Hepatobiliary disorders) | 2 | 0 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 0 | 1
Immune-mediated hepatitis (Hepatobiliary disorders) | 2 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 2 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Abscess limb (Infections and infestations) | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 1 | 0 | 0
Anal abscess (Infections and infestations) | 1 | 2 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
Bacterial diarrhoea (Infections and infestations) | 0 | 1 | 0
Biliary tract infection (Infections and infestations) | 2 | 1 | 2
Bronchitis (Infections and infestations) | 1 | 0 | 0
COVID-19 (Infections and infestations) | 12 | 3 | 2
COVID-19 pneumonia (Infections and infestations) | 1 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 2
Cholangitis infective (Infections and infestations) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Endocarditis (Infections and infestations) | 0 | 0 | 1
Enterocolitis bacterial (Infections and infestations) | 0 | 1 | 0
Eye infection bacterial (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 1
Gastroenteritis clostridial (Infections and infestations) | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Groin abscess (Infections and infestations) | 1 | 0 | 0
Hepatic infection (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 1
Klebsiella sepsis (Infections and infestations) | 1 | 0 | 0
Large intestine infection (Infections and infestations) | 0 | 1 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Periodontitis (Infections and infestations) | 1 | 0 | 0
Peritonitis bacterial (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 7 | 4 | 3
Pneumonia moraxella (Infections and infestations) | 1 | 0 | 0
Salmonella bacteraemia (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 11 | 4 | 2
Septic shock (Infections and infestations) | 1 | 1 | 1
Skin infection (Infections and infestations) | 1 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 7 | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hepatic rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 8 | 2 | 0
Amylase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 9 | 2 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 3 | 0 | 0
Blood thyroid stimulating hormone abnormal (Investigations) | 1 | 0 | 0
Electrocardiogram abnormal (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
Lipase increased (Investigations) | 1 | 0 | 0
Liver function test abnormal (Investigations) | 4 | 0 | 1
Liver function test increased (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0
Transaminases increased (Investigations) | 3 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1
White blood cell count decreased (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 2 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 3 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 38 | 26 | 18
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 2
Tumour rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Brain compression (Nervous system disorders) | 1 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0
Cerebral venous sinus thrombosis (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 3 | 0 | 1
Extrapyramidal disorder (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 12 | 7 | 1
Hypertensive encephalopathy (Nervous system disorders) | 1 | 0 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
Parkinson's disease (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Vertebrobasilar stroke (Nervous system disorders) | 1 | 0 | 0
Acute psychosis (Psychiatric disorders) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 6 | 4 | 4
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 2 | 0 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0/360 | 1/158 | 0/186 — This is a gender-specific adverse event that only affects males. So, the number of At Risk participants only includes the total number of male participants.
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Immune-mediated pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Catheterisation venous (Surgical and medical procedures) | 0 | 1 | 0
Renal stone removal (Surgical and medical procedures) | 1 | 0 | 0
Bleeding varicose vein (Vascular disorders) | 2 | 0 | 0
Embolism (Vascular disorders) | 2 | 0 | 0
Embolism arterial (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 3 | 0 | 0
Hypovolaemic shock (Vascular disorders) | 3 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 1
Venous thrombosis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Arm: Cabozantinib + Atezolizumab (N=429) | Single-Agent Cabozantinib (N=188) | Control Arm: Sorafenib (N=207)
Anaemia (Blood and lymphatic system disorders) | 55 | 23 | 24
Neutropenia (Blood and lymphatic system disorders) | 37 | 16 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 43 | 22 | 11
Hypothyroidism (Endocrine disorders) | 93 | 36 | 9
Abdominal pain (Gastrointestinal disorders) | 68 | 25 | 38
Abdominal pain upper (Gastrointestinal disorders) | 35 | 20 | 17
Ascites (Gastrointestinal disorders) | 54 | 24 | 14
Constipation (Gastrointestinal disorders) | 65 | 33 | 23
Diarrhoea (Gastrointestinal disorders) | 215 | 102 | 98
Dyspepsia (Gastrointestinal disorders) | 24 | 14 | 6
Haemorrhoids (Gastrointestinal disorders) | 13 | 10 | 4
Nausea (Gastrointestinal disorders) | 70 | 40 | 30
Stomatitis (Gastrointestinal disorders) | 40 | 25 | 8
Vomiting (Gastrointestinal disorders) | 45 | 34 | 15
Asthenia (General disorders) | 91 | 34 | 37
Fatigue (General disorders) | 113 | 60 | 36
Mucosal inflammation (General disorders) | 47 | 21 | 12
Oedema peripheral (General disorders) | 53 | 22 | 15
Pyrexia (General disorders) | 51 | 23 | 26
Upper respiratory tract infection (Infections and infestations) | 22 | 5 | 2
Urinary tract infection (Infections and infestations) | 36 | 12 | 6
Alanine aminotransferase increased (Investigations) | 134 | 56 | 24
Amylase increased (Investigations) | 37 | 11 | 10
Aspartate aminotransferase increased (Investigations) | 138 | 61 | 30
Blood alkaline phosphatase increased (Investigations) | 34 | 18 | 13
Blood bilirubin increased (Investigations) | 59 | 27 | 24
Blood lactate dehydrogenase increased (Investigations) | 22 | 9 | 8
Blood thyroid stimulating hormone increased (Investigations) | 22 | 16 | 2
Gamma-glutamyltransferase increased (Investigations) | 34 | 14 | 13
Lipase increased (Investigations) | 45 | 8 | 10
Neutrophil count decreased (Investigations) | 27 | 11 | 2
Platelet count decreased (Investigations) | 59 | 27 | 13
Weight decreased (Investigations) | 82 | 48 | 33
White blood cell count decreased (Investigations) | 16 | 11 | 4
Decreased appetite (Metabolism and nutrition disorders) | 128 | 81 | 43
Hypoalbuminaemia (Metabolism and nutrition disorders) | 41 | 13 | 14
Hypokalaemia (Metabolism and nutrition disorders) | 40 | 12 | 12
Hypomagnesaemia (Metabolism and nutrition disorders) | 26 | 13 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 31 | 14 | 9
Hypophosphataemia (Metabolism and nutrition disorders) | 22 | 10 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 34 | 11 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 29 | 9 | 14
Muscle spasms (Musculoskeletal and connective tissue disorders) | 29 | 10 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 32 | 7 | 4
Dizziness (Nervous system disorders) | 23 | 12 | 7
Dysgeusia (Nervous system disorders) | 39 | 17 | 3
Headache (Nervous system disorders) | 34 | 10 | 7
Insomnia (Psychiatric disorders) | 30 | 10 | 8
Proteinuria (Renal and urinary disorders) | 40 | 19 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 41 | 8 | 14
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 52 | 33 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 31 | 9 | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 22 | 10 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 23 | 12 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 15 | 14 | 31
Dry skin (Skin and subcutaneous tissue disorders) | 38 | 15 | 8
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 185 | 82 | 92
Pruritus (Skin and subcutaneous tissue disorders) | 47 | 12 | 14
Rash (Skin and subcutaneous tissue disorders) | 64 | 29 | 38
Hypertension (Vascular disorders) | 106 | 56 | 39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-01-24): https://cdn.clinicaltrials.gov/large-docs/91/NCT03755791/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-05): https://cdn.clinicaltrials.gov/large-docs/91/NCT03755791/SAP_001.pdf